CLINICAL TRIAL: NCT06336694
Title: Development and Validation of a Deep Learning Radiomics Model With Clinical-radiological Characteristics for the Identification of Occult Peritoneal Metastases in Patients With Pancreatic Ductal Adenocarcinoma
Brief Title: A Deep Learning Radiomics Model for Predicting Occult Peritoneal Metastases of Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Siya Shi, clinical doctor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: SYSUFAH2021-025
Record Dates: First submitted 2023-11-26; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Peritoneum metastases confirmed by pathology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- peritoneal metastases: No intervention had been adminstered during treatment of patients.
  Interventions: Procedure: surgery or diagnostic staging laparoscopy
- without peritoneal metastases: No intervention had been adminstered during treatment of patients.
  Interventions: Procedure: surgery or diagnostic staging laparoscopy

INTERVENTIONS:
Procedure: surgery or diagnostic staging laparoscopy — diagnosis of PDAC with peritoneal examination based on the surgical (for tumors treated with surgery) or diagnostic staging laparoscopy findings (for tumors treated with radiotherapy/chemotherapy)

SUMMARY:
Occult peritoneal metastases (OPM) in patients with pancreatic ductal adenocarcinoma (PDAC) are frequently overlooked during imaging. We aimed to develop and validate a CT-based deep learning-based radiomics (DLR) model with clinical-radiological characteristics to identify OPM in patients with PDAC before treatment.

DETAILED DESCRIPTION:
This retrospective, bicentric study included 302 patients with PDAC (training: n = 167, OPM-positive, n=22; internal test: n = 72, OPM-positive, n=9: external test, n=63, OPM-positive, n=9) who had undergone baseline CT examinations between January 2012 and October 2022. Handcrafted radiomics (HCR) and DLR features of the tumor and HCR features of peritoneum were extracted from CT images. Mutual information and least absolute shrinkage and selection operator algorithms were used for feature selection. A combined model, which incorporated the selected clinical-radiological, HCR, and DLR features, was developed using a logistic regression classifier using data from the training cohort and validated in the test cohorts.

ELIGIBILITY:
Inclusion Criteria:

Patients with suspected pancreatic tumors who underwent contrast enhanced CT and pathological examinations at Center 1 and Center 2 were eligible for inclusion in this study.

Exclusion Criteria:

* (a) pathologically diagnosed PDAC by pathology, (b) time intervals between contrast-enhanced CT and pathology less than 2 weeks; (c) history of pancreatic surgery, (d) history of pancreatic malignancy, and (e) poor CT image quality that undermined peritoneal lesion assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected pancreatic tumors who had undergone contrast-enhanced CT and pathological examinations were screened at Center 1 between January 2012 and October 2022 and Center 2 between January 2014 and October 2021.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
diagnosed with peritoneal metastases | immediately after the surgery
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ting Feng, MD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Shi Siya, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
All data generated for this study were from the authors upon reasonable request.